CLINICAL TRIAL: NCT01290380
Title: An Open-label, Multi-center Study to Evaluate the Effects of ASA404 Alone and in Combination With Taxane-based Chemotherapy on the Pharmacokinetics of Simvastatin, Caffeine, Omeprazole, and Diclofenac in Patients With Advanced Solid Tumor Malignancies
Brief Title: A Study to Evaluate the Effects of ASA404 Alone or in Combination With Taxane-based Chemotherapies on the Pharmacokinetics of Drugs in Patients With Advanced Solid Tumor Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASA404A2111
Record Dates: First submitted 2011-01-26; First posted 2011-02-07 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Solid Tumor Malignancies
Keywords: Solid tumor malignancies,; simvastatin,; caffeine,; omeprazole and diclofenac,; ASA404,; PK data
MeSH Terms: interventions — vadimezan

ARMS (1):
- ASA 404 + standard chemotherapy (Experimental): ASA 404 in combination with in combination with standard chemotherapy (paclitaxel + carboplatin or docetaxel) and a cocktail of caffeine, diclofenac, simvastatin and omeprazole
  Interventions: Drug: ASA404, DMXAA, DXAA

INTERVENTIONS:
Drug: ASA404, DMXAA, DXAA — ASA404 (5,6-dimethylxantheone-4-acetic acid) DMXAA or DXAA

SUMMARY:
The purpose of this study is to evaluate the potential inhibitory effects of ASA404 on CYP1A2, CYP2C9, CYP3A4 and CYP2C19 mediated metabolism on the respective probe drugs caffeine, diclofenac, simvastatin, and omeprazole, respectively. This will be accomplished by the simultaneous administration of four substrates as part of a cocktail in order to characterize the potential for in-vivo drug-drug interactions. This cocktail approach has been proposed per FDA guidance as a screening tool for potential in-vivo drug-drug interactions Compared to the individual administration of specific probes in multiple studies, simultaneous administration of multiple in-vivo probes of drug-metabolizing enzymes offer several distinct advantages such as minimizing the confounding influence of inter-individual and intra-individual variability over time. Substrates for the CYP enzymes were chosen based on the FDA guidance recommendations taking into account that 1. The substrates are specific for the individual CYP enzymes, 2. There are no interactions among these substrates; and 3. The study will be conducted in a sufficient number of subjects.

ELIGIBILITY:
Inclusion Criteria:

Histologically-proven and radiologically-confirmed diagnosis of advanced or metastatic solid tumors for whom treatment with an investigational agent alone or in combination with docetaxel or placlitaxel +carboplatin is appropriate;

* Body Mass Index (BMI) must be within the range of 18-30;
* A minimum of 4 weeks must have elapsed since the last treatment with other cancer therapies, (i.e. endocrine therapy, immunotherapy, chemotherapy, ect);
* Willing and able to remain in the clinic for at least 2 days (the night before dosing and the night after dosing 24 hours) for the 3 x's receiving the cocktail (on Day 1, Day 8 and Day 15 during the

Exclusion Criteria:

* Patients having CNS metastases. (Patients having any clinical signs of CNS metastases must have a CT or MRI of the brain performed to rule out CNS metastases in order to be eligible for the study participation. Patients who have had brain metastases surgically removed or irradiated with no active residual disease confirmed by imaging are allowed)
* Patients who have not recovered from all acute radiotherapy-related toxicities;
* Prior exposure to Vascular Disrupting Agents (VDAs) or other vascular targeting agents
* Right bundle branch block (RBBB), complete left bundle branch block (LBBB), bifascicular block (right bundle branch block with either left anterior hemiblock or left posterior hemiblock)
* Concomitant use of drugs with a risk of QT prolongation and/or causing torsade de pointes

If patient will be treated with paclitaxel:

* Known allergy or hypersensitivity to platinum-containing drugs, taxanes, other drugs formulated in Cremophor EL (polyoxyethylated castor oil) or any known excipients of these drugs
* Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions while taking paclitaxel and therefore are not considered effective contraceptive methods for this study when used as a single agent. Patients taking oral, implantable, or injectable contraceptives who are not willing or otherwise unable to use a concomitant barrier method will be excluded. The Investigator shall counsel the patient accordingly. For a list of substrates of human liver microsomal P450 enzymes, visit website (http://medicine.iupui.edu/flockhart/)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
evaluate the effects of ASA404 on the pharmacokinetics of a cocktail of simvastatin, caffeine, omeprazole, and diclofenac in patients with advanced malignancies. | 12 months
evaluate the effects of ASA404 combined with either paclitaxel + carboplatin or docetaxel on the pharmacokinetics of a cocktail of simvastatin, caffeine, omeprazole, and diclofenac in patients with advanced malignancies. | 12 months

SECONDARY OUTCOMES:
Pharmacokinetic parameters of caffeine, diclofenca, simvastatin, and omeprazole, including AUC (0-tlast), AUC (0-inf), t½,CL/F, Vz/F, Cmax, and tmax. | 12 months
Pharmacokinetic parameters of ASA404 including AUC (0-tlast), Cmax, and Tmax | 4 Months
assessment of safety based mainly on the frequency and severity of adverse events and the number of laboratory values worsening from baseline based on the CTCAE grade. | 4 months
  Other safety data (e.g. vital signs, electrocardiograms, and ophthalmic assessments) will be considered as appropriate.
assess the safety and tolerability of ASA404 | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - The University of Texas Science Center at Houston, Houston, Texas
  - University of Wisconsin & Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin